CLINICAL TRIAL: NCT03915210
Title: Physical Activity Level, Pulmonary Functions and Quality of Life in Candidates of Hematopoietic Stem Cell Transplantation and Healthy Individuals: a Cross-sectional Study
Brief Title: Physical Inactivity in Candidates of HSCT
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Associate professor, Gazi University
Other Study IDs: GaziUniversity18
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Hematopoietic Stem Cell Transplantation
Keywords: Energy metabolism; Exercise; respiratory function test; quality of life; leisure activities; hematopoietic stem cell transplantation
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Candidates of HSCT: Physical activity level using a metabolic holter device, dynamic lung volumes (FEV1, FVC, FEV1/FVC, PEF, FEF25-75%) using a spirometer and quality of life using European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 version 3.0 were objectively evaluated.
- Healthy individuals: Physical activity level using a metabolic holter device, dynamic lung volumes (FEV1, FVC, FEV1/FVC, PEF, FEF25-75%) using a spirometer and quality of life using European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 version 3.0 were objectively evaluated.

SUMMARY:
Decreased number of steps and poorer quality of life are prevalently observed among candidates of hematopoietic stem cell transplantation (HSCT). However, impairments in other aspects of physical activity measurement including energy expenditure, physical activity duration, metabolic equivalents of daily task (METs) and lying down duration are still unknown in candidates based on comparison with healthy individuals, which was therefore aimed to investigate in current study.

DETAILED DESCRIPTION:
In recent years, hematopoietic stem cell transplantation (HSCT) has been largely used to cure not only many hematologic malignancies but also autoimmune diseases and even genetic diseases. Advances in the HSCT and other cancer treatment approaches including supportive care practices provide patients better survival time nowadays. However, as life expectancy for recipients is increasing up to 85% for being alive 10 years after HSCT, post-HSCT complications are concurrently increasing. After HSCT, recipients may suffer from many infectious complications, cytopenia, immunosuppression, graft versus host disease, a lot of organ involvements and even secondary malignancies. In addition, they are also exposed to immobility condition, physical inactivity, depressive symptoms, psychosocial distress, fatigue, and complications of musculoskeletal, respiratory and cardiovascular systems rely on mostly treatments and treatment related with complications all of which have a negative impact on the survival, physical functions and quality of life of recipients. Hence, the guidelines recommend to all recipients both routine evaluations of clinical and cardiovascular risk factors, and also complying with healthy life style including doing regular physical activity and exercises.

On the other hand, chemotherapy, radiation therapy and further conditioning regimens are required to exterminate the abnormally proliferating cancer cells in patients with hematologic malignancies before HSCT, which also leads to pre-HSCT complications. These complications are observed as physical inactivity, abnormal pulmonary functions, muscle weakness, decreased exercise capacity, evident fatigue, psychological mood disorders and poorer quality of life in these patients until HSCT. Should immobility and physical inactivity extend, the patients may need to respiratory support including oxygen supply, noninvasive or invasive mechanic ventilation. As previously shown, these impairments especially physical inactivity have even existed in patients with hematologic malignancies at the period of pre-diagnosis and early diagnosis. While 33.8% of patients (n=438) could achieve the daily/weekly exercise criteria of guidelines during the time of pre-diagnosis, only 6.5% of patients could perform physical activity during anticancer treatments. In that study, physical activity level was evaluated using a questionnaire, and the patients meeting public health exercise guidelines have reported higher quality of life level. According to results of another study with higher sample size (n=3060), 1392 (46%) of patients are physically active based on their responses to questions at the pre-diagnosis period. However, the most striking result to emerge from the data in 2018 is that these active patients have considerably higher survival rates rather than insufficiently active patients. As demonstrated in 2014 (n=29), 61% of patients with early diagnosis meet the physical activity guidelines, and patients walk about 6.149 steps/d before the start of chemotherapy which was evaluated via a tri-axial accelerometer. As known, although patients have survived after HSCT, these problems have not meliorated in survivors over a long time after HSCT. Therefore, guidelines recommend that the patients should be oriented for rehabilitation in order to maximize muscle strength, functional mobility and quality of life of patients before the patients are subject to the process of HSCT.

Evaluation and counseling of physical activity have become one of the most challenging topics recently; however, there is confusion in the meaning and usage of this term. Original definition of physical activity is "Physical activity is defined as any bodily movement produced by skeletal muscles that results in energy expenditure. Physical activity in daily life can be categorized into occupational, sports, conditioning, household, or other activities. Exercise is a subset of physical activity that is planned, structured, and repetitive and has as a final or an intermediate objective the improvement or maintenance of physical fitness.". In the literature, researchers have mostly tend to only one aspect of physical activity measurement in candidates of HSCT which is either steps count or estimation of physical activity intensity as regard to metabolic equivalent of daily task (MET). In fact, reason of this situation was that less objective tools such as questionnaire, questions, and pedometers were used to evaluate physical activity level in candidates. There is just a few studies used an objective device like triaxial accelerometer in the literature.

Physical inactivity as a cardiovascular risk factor is related with higher risks of cardiovascular diseases and complications after HSCT. Therefore, it is important to assess detailed physical activity along with its all aspects including energy expenditure, number of steps, activity types and durations in candidates of HSCT. However, impairments in energy expenditure, physical activity duration, metabolic equivalents of daily task (METs) and lying down duration are still unknown in candidates versus healthy individuals who are age and gender matched counterparts of candidates. Hence, it was aimed to compare physical activity parameters, pulmonary functions and quality of life scores of candidates with healthy individuals in the current study.

ELIGIBILITY:
Inclusion Criteria for the candidates:

* being aged between 18 and 65 years, being a candidate for either allogeneic or autologous HSCT before the start of conditioning regimen who were orientated from Bone Marrow Transplantation Unit,
* having a diagnosis with a hematologic malignancy,
* being clinically stabile,
* being functionally mobile
* receiving optimal standard medical therapy including antibiotics, supplements and other drugs.

Exclusion Criteria for the candidates:

* having cooperation problems, having orthopedic or neurological disease with a potential to limit daily walking,
* having comorbidities such as chronic obstructive pulmonary disease, cardiac diseases, acute infections and/or active hemorrhage (with hemoglobin values ≤8 g/L and platelet count ≤10.000 mm3)

Inclusion Criteria for the healthy individuals:

* being eager to participate to the study
* being aged between 18 and 65 years,

Exclusion Criteria for the healthy individuals:

* having any diagnosis of chronic diseases
* being current smokers
* being ex-smokers (≥10 pack*years)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients were previously diagnosed with a hematological malignancy and determined to be a candidate for allogeneic-HSCT who were orientated from Bone Marrow Transplantation Unit for rehabilitation program. Healthy individuals were recruited from staff in the university and their healthy relatives.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Physical activity measurement | during a total of 48 hours
  Physical activity levels of all participants were assessed with a metabolic holter device.

SECONDARY OUTCOMES:
Evaluation of dynamic lung volumes | 5 minutes
  To assess dynamic lung volumes involving forced vital capacity (FVC), forced expiratory volume in one second (FEV1), forced expiratory volume in one second/forced vital capacity (FEV1/FVC), peak expiratory flow (PEF) and forced expiratory flow at 25%-75% (FEF25-75%), a spirometer was used. Guidelines were taken reference for this measurement. These values were recorded as percentages of predicted values.
General quality of life assesment: European Organization for Research and Treatment of Cancer QOL Questionnaire (EORTCQOL) | 2 minutes
  European Organization for Research and Treatment of Cancer QOL Questionnaire C30 version3.0 was used to evaluate quality of life impairment. This is a self-administered questionnaire which consists of five functional subscales along with a social functioning subscale, three symptom subscales with also a fatigue subscale, a global health status subscale, and several single items. All item scores are converted to values from 0 to 100. Higher values show higher health levels in functional and social functioning subscales, a higher quality of life level in global health status subscale, and increased presence of symptoms in both symptom and fatigue subscales.

CONTACTS AND LOCATIONS:
Overall Officials: Gülşah Barğı, PhD, Study Chair — Gazi University; Meral Boşnak Güçlü, PhD, Study Director — Gazi University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Copelan EA. Hematopoietic stem-cell transplantation. N Engl J Med. 2006 Apr 27;354(17):1813-26. doi: 10.1056/NEJMra052638. No abstract available. PMID 16641398
- [Result] Paudel N, Schulze D, Gentzler RD, Evens AM, Helenowski I, Dillehay G, Frankfurt O, Mehta J, Donnelly ED, Gordon LI, Winter JN, Mittal BB. Patterns of Failure and Survival Outcomes after Total Lymphoid Irradiation and High-Dose Chemotherapy with Autologous Stem Cell Transplantation for Relapsed or Refractory Classical Hodgkin Lymphoma. Int J Radiat Oncol Biol Phys. 2019 Jun 1;104(2):436-446. doi: 10.1016/j.ijrobp.2019.02.007. Epub 2019 Feb 11. PMID 30763660
- [Result] Mohammed J, Smith SR, Burns L, Basak G, Aljurf M, Savani BN, Schoemans H, Peric Z, Chaudhri NA, Chigbo N, Alfred A, Bakhsh H, Salooja N, Chris Chim A, Hashmi SK. Role of Physical Therapy before and after Hematopoietic Stem Cell Transplantation: White Paper Report. Biol Blood Marrow Transplant. 2019 Jun;25(6):e191-e198. doi: 10.1016/j.bbmt.2019.01.018. Epub 2019 Jan 15. PMID 30658224
- [Result] Wingard JR, Majhail NS, Brazauskas R, Wang Z, Sobocinski KA, Jacobsohn D, Sorror ML, Horowitz MM, Bolwell B, Rizzo JD, Socie G. Long-term survival and late deaths after allogeneic hematopoietic cell transplantation. J Clin Oncol. 2011 Jun 1;29(16):2230-9. doi: 10.1200/JCO.2010.33.7212. Epub 2011 Apr 4. PMID 21464398
- [Result] Majhail NS, Rizzo JD, Lee SJ, Aljurf M, Atsuta Y, Bonfim C, Burns LJ, Chaudhri N, Davies S, Okamoto S, Seber A, Socie G, Szer J, Van Lint MT, Wingard JR, Tichelli A; Center for International Blood and Marrow Transplant Research (CIBMTR); American Society for Blood and Marrow Transplantation (ASBMT); European Group for Blood and Marrow Transplantation (EBMT); Asia-Pacific Blood and Marrow Transplantation Group (APBMT); Bone Marrow Transplantation Society of Australia and New Zeland (BMTSANZ); East Mediterrnean Blood and Marrow Transplantation Group (EMBMT); Sociedale Brasileira de Transplante de Medula Ossea (SBTMO). [Recommended screening and preventive practices for long-term survivors after hematopoietic cell transplantation]. Rinsho Ketsueki. 2014 Jun;55(6):607-32. Japanese. PMID 24975331
- [Result] Vermaete N, Wolter P, Verhoef G, Gosselink R. Physical activity and physical fitness in lymphoma patients before, during, and after chemotherapy: a prospective longitudinal study. Ann Hematol. 2014 Mar;93(3):411-24. doi: 10.1007/s00277-013-1881-3. Epub 2013 Aug 21. PMID 23963412
- [Result] Hung YC, Bauer J, Horsley P, Waterhouse M, Bashford J, Isenring E. Changes in nutritional status, body composition, quality of life, and physical activity levels of cancer patients undergoing autologous peripheral blood stem cell transplantation. Support Care Cancer. 2013 Jun;21(6):1579-86. doi: 10.1007/s00520-012-1698-y. Epub 2013 Jan 10. PMID 23306934
- [Result] White AC, Terrin N, Miller KB, Ryan HF. Impaired respiratory and skeletal muscle strength in patients prior to hematopoietic stem-cell transplantation. Chest. 2005 Jul;128(1):145-52. doi: 10.1378/chest.128.1.145. PMID 16002928
- [Result] Morishita S, Kaida K, Yamauchi S, Wakasugi T, Ikegame K, Ogawa H, Domen K. Relationship of physical activity with physical function and health-related quality of life in patients having undergone allogeneic haematopoietic stem-cell transplantation. Eur J Cancer Care (Engl). 2017 Jul;26(4). doi: 10.1111/ecc.12669. Epub 2017 Feb 21. PMID 28220548
- [Result] Morishita S, Kaida K, Tanaka T, Itani Y, Ikegame K, Okada M, Ishii S, Kodama N, Ogawa H, Domen K. Prevalence of sarcopenia and relevance of body composition, physiological function, fatigue, and health-related quality of life in patients before allogeneic hematopoietic stem cell transplantation. Support Care Cancer. 2012 Dec;20(12):3161-8. doi: 10.1007/s00520-012-1460-5. Epub 2012 Apr 12. PMID 22526152